CLINICAL TRIAL: NCT04423536
Title: Predictive Value of a SNP Signature and Liquid Biopsy in Natural Killer T-cell Lymphoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Qingqing Cai, Chief physician, Sun Yat-sen University
Other Study IDs: B2020-035
Record Dates: First submitted 2020-06-07; First posted 2020-06-09 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2022-05

CONDITIONS: Natural Killer T-cell Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- tested group
- controlled group

SUMMARY:
The purpose of this study is to determine the Predictive value of a SNP signature and liquid biopsy in patients with natural killer T-cell lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* biopsy proved Natural Killer T-cell Lymphoma
* newly diagnosed patients

Exclusion Criteria:

* patients with biopsy samples unavailable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adults
Sampling Method: Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2021-03-09 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 5-years

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen Universitiy Cancer Center, Sun Yat-Sen University,, Guangzhou, China